CLINICAL TRIAL: NCT02556671
Title: Platelet Reactivity Over Time After Receiving Clopidogrel Among Moderate CKD Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Platelet Reactivity After Receiving Clopidogrel Among Moderate CKD Patients Undergoing PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruqiong Nie (Other)
Responsible Party: Sponsor-Investigator, Ruqiong Nie, director of cardiology, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Other Study IDs: SunYatsenU2H
Record Dates: First submitted 2015-08-27; First posted 2015-09-22 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Moderate CKD Patients Undergoing PCI
- Normal renal function Patients Undergoing PCI

SUMMARY:
Dual antiplatelet therapy (DAPT) with standard doses of aspirin and clopidogrel has long been the cornerstone in patients undergoing percutaneous coronary intervention (PCI). However, inhibition of platelet activation and aggregation after DAPT varies greatly among patients. Some clinical studies have demonstrated that patients with high on-treatment platelet reactivity are at increased risk of major adverse cardiovascular events. Tailored antiplatelet therapy seems offer an opportunity to improve outcomes after coronary stenting by drug adjustment based on platelet function testing. Unfortunately, the results of 3 major prospective trials (GRAVITAS, ARCTIC, TRIGGER PCI) of personalized antiplatelet therapy are neutral. In these studies, platelet function was only assessed by a single measurement and a single method early after the start of antiplatelet treatment. To test the stability of platelet reactivity measurements over time among patients undergoing PCI, investigators use 3 methods (VerifyNow P2Y12 assay, Flow cytometric assessment of the phosphorylation status of VASP, light transmittance aggregometry) for platelet function testing in 2 periods (~14days), with maintenance doses of clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old.

2.15 ≤ eGFR < 60 ml/min/1.73 m2.

3. Clinically stable and following PCI between 4 weeks and 1 year.

4. On clopidogrel (75mg/d) and aspirin (100mg/d) treatment at least 4 weeks.

Exclusion Criteria:

1. Conditions that alter platelet function.
2. Conditions that increase bleeding risk.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dual antiplatelet therapy (DAPT) with standard doses of aspirin and clopidogrel has long been the cornerstone in patients undergoing percutaneous coronary intervention (PCI). However, inhibition of platelet activation and aggregation after In these studies, platelet function was only assessed by a single measurement and a single method early after the start of antiplatelet treatment. To test the stability of platelet reactivity measurements over time among patients undergoing PCI, we use 3 methods (VerifyNow P2Y12 assay, Flow cytometric assessment of the phosphorylation status of VASP, light transmittance aggregometry) for platelet function testing in 2 periods (~14days), with maintenance doses of clopidogrel.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Individual Platelet Reactivity Measured by VerifyNow P2Y12 Assay Over Time after Receiving Clopidogrel among Moderate CKD Patients Undergoing Percutaneous Coronary Intervention -- A Cross-Sectional Study | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ruqiong nie, Study Chair — Sunyatsen memorial hospital
Locations (1):
- Sunyatsen memorial hospital, Guangzhou, China